CLINICAL TRIAL: NCT05579379
Title: DESENSITIZE-PD: Intestinal Levodopa + Entacapone Therapy (Lecigon®) to Support Dopaminergic Desensitization in Parkinson's Disease
Brief Title: DESENSITIZE-PD: Intestinal Levodopa + Entacapone Therapy (Lecigon®) to Support Dopaminergic Desensitization in PD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: STADAPHARM GmbH (Unknown)
Responsible Party: Principal Investigator, Daniel Weiss, Prof. Dr., University Hospital Tuebingen
Other Study IDs: 388/2022BO2
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; dopaminergic sensitization; hyperdopaminergic complications; neuropsychiatric complications; intestinal L-Dopa therapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
20 patients with idiopathic Parkinson's disease, who are planned to undergo intestinal L-Dopa + entacapone (Lecigon®) treatment will be included into this observational single-armed study. These patient will be observed for hyperdopaminergic complications and neuropsychiatric fluctuations postprocedure at 3, 6 and 12 months.

DETAILED DESCRIPTION:
This study is planned as non-interventional observational single-armed study in patients that are planned to undergo intestinal L-Dopa + entacapone (Lecigon®) treatment as regular treatment choice outside the study protocol and under the accepted regulatory approval and indication criteria (according to German "Fachinformation Lecigon®"). Patients will be observed at the pre-interventional baseline (oral treatment, before treatment initiation with Lecigon®), 3-month, 6-month follow-up, and final 12-month follow-up. As primary interest, the investigator will analyze the contrast of the pre-interventional baseline and 12-month follow-up in terms of the Ardouin Behavioural Scale which evaluates the hyperdopaminergic complications and neuropsychiatric fluctuations in a semi-structured interview. As additional exploratory outcomes, the investigator will study the "Neuropsychiatric fluctuation scale", impulse control disorders with the "QUIP rating scale (QUIP-RS)". Moreover, the investigator will study apathy outcomes using the "Apathy Evaluation Scale" that mainly relates to the dopaminergic off-state. Outcomes of post-interventional apathy are particularly important, since i) they may coincide with hypodopaminergic off-states, and ii) since outcomes of postoperative apathy are a limitation of existing DBS therapy. Avoiding worsening of apathy might be a strength of intestinal L-Dopa therapy in this regard. Further, the investigator will study established measures of motor sensitization/de-sensitization in particular motor fluctuations and dyskinesia (MDS-UPDRS IV) and Unified Dyskinesia Rating Scale (UDysRS). For completeness, the investigator will characterize MDS-UPDRS III motor state in addition.

Since dopaminergic desensitization occurs with considerable delay of rather weeks and months after changing oral to continuous treatment, the investigator expect a reduction of dopaminergic motor and neuropsychiatric complications within the first 6 months from introducing Lecigon® together with a stable course until final 12-month follow-up. The outcomes will be decided as contrast of the pre-interventional baseline (V0) in best oral treatment compared to 12 month follow-up of Lecigon® treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written declaration of consent
* Age > 18 years and < 80 years
* Idiopathic Parkinson's syndrome (according to British Brain Bank criteria), including genetic forms
* L-dopa responsive Parkinson's syndrome
* Duration of disease > 5 years
* The treatment decision for Lecigon® was made as a regular treatment decision according to the established indication criteria outside the study
* Motor fluctuations on oral dopaminergic therapy with uncontrolled motor off symptoms
* Presence or history of dyskinesia based on available medical records or self-reported history
* History of dopaminergic neuropsychiatric therapy complications based on available physician's letters or self-reported history:

  * impulse control disorders or
  * dopamine dysregulation syndrome or
  * off-condition apathy or
  * affective response fluctuations or
  * affective hypomanic or manic complications
  * hyperdopaminergic behavioral complications (such as binge eating or hobbyism or punding or increased creativity or risk seeking behavior; analogous to Ardouin Behaviour Scale Chapter IV - hyperdopaminergic behaviors).

Exclusion Criteria:

* Dementia according to ICD-10 criteria; mild cognitive impairment (MCI) according to screening tools such as MoCA or MMSE is not considered an exclusion criterion as long as ICD-10 criteria for dementia are not met regardless of MoCA/MMSE score.
* Acute paranoid psychosis or suicidality (however, impulse control disorder or dopamine dysregulation syndrome is not an exclusion criterion; illusions or (pseudo)-hallucinations are also not an exclusion criterion, as long as there is no risk to the patient or others according to clinical judgment; patients may be allowed to participate in the study after remission of the psychosis/suicidality)
* Pregnancy
* Contraindications to therapy with Lecigon® according the Summary of Product Characteristics (SmPC)

  * Hypersensitivity to the active ingredients of Lecigon®.
  * Narrow-angle glaucoma
  * Severe heart failure
  * Severe cardiac arrhythmia
  * Acute stroke
  * Severe impairment of liver function
  * Non-selective MAO inhibitors and selective type A MAO inhibitors must not be used concomitantly with Lecigon®. These inhibitors must have been discontinued at least two weeks prior to starting treatment with Lecigon®. Lecigon® may be used concomitantly with the manufacturer's recommended dose of an MAO inhibitor with selectivity for MAO type B (e.g., selegiline hydrochloride)
  * Conditions in which sympathomimetics (adrenergics) are contraindicated, e.g., pheochromocytoma, hyperthyroidism, and Cushing's syndrome.
  * Previous malignant neuroleptic syndrome (NMS) and/or nontraumatic rhabdomyolysis.
  * Suspected undiagnosed skin lesions or history of melanoma (levodopa could activate malignant melanoma).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll patients with Parkinson's disease, who are eligible for intestinal treatment with Lecigon® as a regular treatment option outside of the study protocol and under the accepted eligibility and indication criteria.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Ardouin Behavioural Scale | At baseline, 3 months, 6 months and 12 months, respectively
  To evaluate the hyperdopaminergic complications and neuropsychiatric fluctuations from baseline to 12-months follow-up.
  Minimum value: 0, maximum value: 84, higher score means worse outcome.

SECONDARY OUTCOMES:
Neuropsychiatric Fluctuation Scale | At baseline, 3 months, 6 months and 12 months, respectively
  To identify and quantify neuropsychiatric fluctuations during motor fluctuations.
  Minimum value for OFF items: 0, maximum value for OFF items: 30, higher score means worse outcome.
  Minimum value for ON items: 0, maximum value for ON items: 30, higher score means worse outcome.
Questionnaire for impulsive-compulsive disorders in Parkinson's disease (QUIP) | At baseline, 3 months, 6 months and 12 months, respectively
  To assess the severity of impulsive-compulsive disorders. Minimum value: 0, maximum value: 112, higher score means worse outcome.
Apathy Evaluation Scale | At baseline, 3 months, 6 months and 12 months, respectively
  To quantify and characterize the apathy. Minimum value: 0, maximum value: 54, higher score means worse outcome.
Movement Disorders Society -Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III | At baseline, 3 months, 6 months and 12 months, respectively
  To measure the severity of Parkinson symptoms. Minimum value: 0, maximum value: 132, higher score means worse outcome.
Movement Disorders Society -Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part IV | At baseline, 3 months, 6 months and 12 months, respectively
  To measure the severity of motor complications. Minimum value: 0, maximum value: 24, higher score means worse outcome.
Unified Dyskinesia Rating Scale (UDyRS) | At baseline, 3 months, 6 months and 12 months, respectively
  To evaluate involuntary movements. Minimum value: 0, maximum value: 104, higher score means worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Weiss, MD, Principal Investigator — University Hospital Tuebingen

IPD SHARING:
Plan to Share IPD: Undecided
A study database will be established with our Institute for Clinical Epidemiology and Applied Biometry. Pseudonymized data can be made available after publication upon reasonable request to the Principal Investigator

REFERENCES:
- [Background] Weiss D, Volkmann J, Fasano A, Kuhn A, Krack P, Deuschl G. Changing Gears - DBS For Dopaminergic Desensitization in Parkinson's Disease? Ann Neurol. 2021 Nov;90(5):699-710. doi: 10.1002/ana.26164. Epub 2021 Jul 20. PMID 34235776
- [Background] Weiss D, Ebersbach G, Moller JC, Schwarz J, Arlt C, Fritz B, Sensken SC, Eggert K. Do we start too late? Insights from the real-world non-interventional BALANCE study on the present use of levodopa/carbidopa intestinal gel in advanced Parkinson's disease in Germany and Switzerland. Parkinsonism Relat Disord. 2022 Oct;103:85-91. doi: 10.1016/j.parkreldis.2022.08.018. Epub 2022 Aug 24. PMID 36087571
- [Background] Schmitt E, Krack P, Castrioto A, Klinger H, Bichon A, Lhommee E, Pelissier P, Fraix V, Thobois S, Moro E, Martinez-Martin P. The Neuropsychiatric Fluctuations Scale for Parkinson's Disease: A Pilot Study. Mov Disord Clin Pract. 2018 Mar 23;5(3):265-272. doi: 10.1002/mdc3.12607. eCollection 2018 May-Jun. PMID 30363450
- [Background] Papay K, Mamikonyan E, Siderowf AD, Duda JE, Lyons KE, Pahwa R, Driver-Dunckley ED, Adler CH, Weintraub D. Patient versus informant reporting of ICD symptoms in Parkinson's disease using the QUIP: validity and variability. Parkinsonism Relat Disord. 2011 Mar;17(3):153-5. doi: 10.1016/j.parkreldis.2010.11.015. Epub 2010 Dec 24. PMID 21186135
- [Background] Probst CC, Winter LM, Moller B, Weber H, Weintraub D, Witt K, Deuschl G, Katzenschlager R, van Eimeren T. Validation of the questionnaire for impulsive-compulsive disorders in Parkinson's disease (QUIP) and the QUIP-rating scale in a German speaking sample. J Neurol. 2014 May;261(5):936-42. doi: 10.1007/s00415-014-7299-6. Epub 2014 Mar 9. PMID 24609972
- [Background] Weintraub D, Mamikonyan E, Papay K, Shea JA, Xie SX, Siderowf A. Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale. Mov Disord. 2012 Feb;27(2):242-7. doi: 10.1002/mds.24023. Epub 2011 Dec 1. PMID 22134954